CLINICAL TRIAL: NCT01866124
Title: MAM'Out Project - Evaluation of Multiannual and Seasonal Cash Transfers to Prevent Acute Malnutrition
Acronym: MAM'Out
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Action Contre la Faim (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University Ghent (Other); AgroParisTech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACF0213; 1U01GH000646-01 (NIH)
Record Dates: First submitted 2013-05-07; First posted 2013-05-31 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Acute Malnutrition
Keywords: acute malnutrition; multiannual and seasonal cash transfers; safety nets; Burkina Faso

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cash transfer (Experimental): Mothers are the primary recipient of the CT. The proposed approach will be based on monthly seasonal CTs during 5 months, from May to September, for two years (2013 and 2014). A monthly 10 000 FCFA will be transferred to the selected households.
  These CTs will be done via mobile phones, in collaboration with the mobile phone company Airtel.
  Interventions: Other: Cash transfer
- Comparison group (No Intervention)

INTERVENTIONS:
Other: Cash transfer — Recipient of transfers Mothers are the primary recipient of the CT. Cash is transferred using mobile phone credits that can be cashed at specific cash points provided by a telecom company.
  Other Names: Multiannual and seasonal cash transfer
  Arms: Cash transfer

SUMMARY:
The MAM'Out research project aims at evaluating a seasonal and multi-annual cash transfer program in the framework of a safety net to prevent acute malnutrition by children under 24 months, in terms of effectiveness and cost-effectiveness in the Tapoa province (East region of Burkina Faso, Africa). The program will be targeted to economically vulnerable households with children less than 1 year old at the time of inclusion and the cash distributed to mothers. The transfers will be assimilated to unconditional ones, leading to beneficiaries' self-determination on the use that will be made of cash. This study will be designed as a two-arm cluster randomized intervention trial, based on randomization of rural villages of the Tapoa province. One arm will receive the intervention and one will be a control arm. The main outcomes will be the cumulative incidence of acute malnutrition (or wasting) and the cost-effectiveness. Anthropometric measures (height, weight and MUAC) will be measured, as well as indicators of dietary diversity, food security, health center frequentation, families' expenses and morbidities. Questionnaires and 24-hour food recalls will also be analyzed. Finally, based on a model theory framework built a priori, the pathways used by the cash to have an effect on the prevention of under-nutrition will be assessed.

DETAILED DESCRIPTION:
At international level, the WHO formulated guidelines for the treatment of severe acute malnutrition (or wasting) (WHO 1999, and more recently ACF 2011), and guidelines for moderate acute malnutrition (or wasting) are in the process of formulation. In contrast, surprisingly little is known on preventive schemes for acute malnutrition. In Haiti, Ruel et al (2008) found that targeting nutrition interventions to prevent children from becoming malnourished might be more effective than curative treatment to reduce child wasting. In addition, recent preventive trials in humanitarian settings focused on the use of food-based strategies, especially ready-to-use food (Isanaka, 2009; Hendricks, 2010; Parikh, 2010; Imbad, 2011; Huybregts, 2012). However, it is well known that the causes of under-nutrition are numerous and also relate to inadequate health and care practices, lack of food diversification, food insecurity… Therefore, the MAM'Out research project aims at assessing a context-adapted preventive approach, which is likely to influence several underlying causes of under-nutrition and not based primarily on food supplementation. The objective is to provide an evidence base for this alternative approach, in order that proven intervention be taken into account for scale-up at policy-making levels.

ELIGIBILITY:
Inclusion Criteria:

* Poor or very poor household (HEA criteria)
* Having at least one children under 1 year old at the time of inclusion

Exclusion Criteria:

* Medium or rich economic status (HEA criteria)
* no child under one year old at the time of inclusion
* not living in one of the 32 selected villages in the Tapoa province

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1278 (Actual)
Dates: Start 2013-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of child wasting | 3-monthly until 24 months after inclusion
  Record of the child's height, weight to compute Weight for Height Z-scores (WHZ scores) (wasting defined as WHZ<-2 or Edema)
Incremental cost-effectiveness ratio | 24 months after inclusion
  Calculation of a cost-effectiveness ratio at the end of the study

SECONDARY OUTCOMES:
cumulative incidence of the state of stunting | 3-monthly until 24 months after inclusion
mean height-for-age Z-score | 3-monthly until 24 months after inclusion
mean weight-for-length Z-score | 3-monthly until 24 months after inclusion
mid-upper arm circumference (MUAC) | 3-monthly until 24 months after inclusion
edema | 3-monthly until 24 months after inclusion
Prevalence of diarrhea | 3-monthly until 24 months after inclusion
Prevalence of acute respiratory infections | 3-monthly until 24 months after inclusion
Reported measle | 3-monthly until 24 months after inclusion
  the symptoms used to detect measles will be the following ones (from WHO) : tiny white spots on the inside of the mouth and rash on the face and/or the body

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kolsteren, MD, PhD, Principal Investigator — Universiteit Gent, Institute of Tropical Medicine of Antwerp (Belgium); Myriam Ait Aissa, MSc, Study Director — Action Contre la Faim
Locations (1):
- Action Contre la Faim - Burkina Faso, Diapaga, Tapoa, Burkina Faso

REFERENCES:
- [Derived] Tonguet-Papucci A, Houngbe F, Huybregts L, Ait-Aissa M, Altare C, Kolsteren P, Huneau JF. Unconditional Seasonal Cash Transfer Increases Intake of High-Nutritional-Value Foods in Young Burkinabe Children: Results of 24-Hour Dietary Recall Surveys within the Moderate Acute Malnutrition Out (MAM'Out) Randomized Controlled Trial. J Nutr. 2017 Jul;147(7):1418-1425. doi: 10.3945/jn.116.244517. Epub 2017 May 31. PMID 28566529
- [Derived] Tonguet-Papucci A, Houngbe F, Lompo P, Yameogo WME, Huneau JF, Ait Aissa M, Kolsteren P. Beneficiaries' perceptions and reported use of unconditional cash transfers intended to prevent acute malnutrition in children in poor rural communities in Burkina Faso: qualitative results from the MAM'Out randomized controlled trial. BMC Public Health. 2017 May 30;17(1):527. doi: 10.1186/s12889-017-4453-y. PMID 28558709
- [Derived] Houngbe F, Tonguet-Papucci A, Altare C, Ait-Aissa M, Huneau JF, Huybregts L, Kolsteren P. Unconditional Cash Transfers Do Not Prevent Children's Undernutrition in the Moderate Acute Malnutrition Out (MAM'Out) Cluster-Randomized Controlled Trial in Rural Burkina Faso. J Nutr. 2017 Jul;147(7):1410-1417. doi: 10.3945/jn.117.247858. Epub 2017 May 24. PMID 28539413
- [Derived] Tonguet-Papucci A, Huybregts L, Ait Aissa M, Huneau JF, Kolsteren P. The MAM'Out project: a randomized controlled trial to assess multiannual and seasonal cash transfers for the prevention of acute malnutrition in children under 36 months in Burkina Faso. BMC Public Health. 2015 Aug 8;15:762. doi: 10.1186/s12889-015-2060-3. PMID 26253152